CLINICAL TRIAL: NCT04404621
Title: Computer Presented and Physical Exercises to Maintain Cognitive Function and Emotional Health in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2000026437
Record Dates: First submitted 2020-05-22; First posted 2020-05-27 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Cognitive Function; Depression in Old Age
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cross-Over Sequence A (Experimental): Participants in this arm will be randomized to receive the 18 week program first and be in treatment as usual comparison condition in the following 18 weeks.
  Interventions: Behavioral: Physical exercise (PE) training and computer-based brain (CBB)
- Cross-Over Sequence B (Experimental): Participants in this arm will be randomized to remain in treatment as usual during the first 18 week period and then receive the 18 week program during the following 18 weeks.
  Interventions: Behavioral: Physical exercise (PE) training and computer-based brain (CBB)

INTERVENTIONS:
Behavioral: Physical exercise (PE) training and computer-based brain (CBB) — 18 weeks of PE and CBB.

SUMMARY:
The aim of this study is to investigate and compare how 18-weeks of computer-based brain training and physical exercise together can improve physical performance, cognitive function and mood in older adults in a cross-over design with participants randomized to receive the intervention first and then be assessed before and after an 18 week period without intervention, or the reverse sequence.

DETAILED DESCRIPTION:
The aim of this study is to investigate and compare how 18-weeks of computer-based brain training and physical exercise together can improve physical performance, cognitive function and mood in older adults in a cross-over design with participants randomized to receive the intervention first and then be assessed before and after an 18 week period without intervention, or the reverse sequence. 80 adults between the ages of 65 and 105 years old will be invited to participate. After providing informed consent, in the case of subjects who are living on units for individuals with memory or other cognitive compromise, after assent from the individual and approval from facility staff, subjects will be randomly assigned to either receive the intervention for 18 weeks and then be followed for an additional 18 weeks, or to be followed for 18 weeks without intervention and then do the intervention for 18 weeks. The intervention will consist of 18 weeks of 60-minute PE sessions 3-4 times/week and 25-minute CBB training sessions 3-4 times a week.

There will be 3 assessments of participants: before and after the first 18-week period and then again after the second 18-week period. Assessments will be done in 2 sessions over a total of 90 minutes and will include demographic, health, physical activity and social activity questionnaires as well as the self-report measures of cognitive function, emotional state and weekly activities; quantitative assessments of physical balance, strength, flexibility blood pressure and heart rate; and tests of cognitive function. Subject medications will be recorded at each assessment. The wait-list control group will receive the same assessments at the same time points.

ELIGIBILITY:
Inclusion Criteria:

* Associated with Whitney center as residents or participants in non-resident programs.
* Able to understand and read English.

Exclusion Criteria:

* Not able to sit in a chair independently.
* Not able to move both arms in simple movement sequence.
* Hearing and vision insufficient to do the computer exercises or follow the PE instructions.
* Not able to remember 3 movements in succession.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-09-12 (Actual); Study Completion 2020-09-12 (Actual)

PRIMARY OUTCOMES:
Composite cognition score | 18 weeks
  Composite from: Flanker Test of Attention; Go/No-Go Test of Response Inhibition; List Sort Working Memory Test; Logical Memory Story Recall; Digit symbol coding; Digit Span Forwards and Backwards; Hopkin's Verbal Learning Test; Trail Making B; Stroop Color Word; Category Verbal Fluency; Reaction Time.
  A composite score will be calculated for each participant at baseline and after training and waitlist periods by first determining Z-scores for each test for each participant at each time point based on means and standard deviations for the entire sample at baseline, and then averaging the individual's Z-scores at that time point.
Sit to Stand in one-minute | 18 weeks
  Number of times able to go from sit to stand in in one minute
Balance - stand on one foot at a time | 18 weeks
  Stand on one foot with the toe of the other foot touching the calf of the standing leg - number of seconds able to maintain. The sum of right and leg foot will be added.
Mood and Quality of Life | 18 weeks
  Composite score from WHODAS, DEMQ QLI and Beck Depression Inventory.
  A composite score will be calculated for each participant at baseline and after training and waitlist periods by first determining Z-scores for total score on each questionnaire for each participant at each time point based on means and standard deviations for the entire sample at baseline, and then averaging the individual's Z-scores at that time point.

SECONDARY OUTCOMES:
Attention and Speed of Processing | 18 weeks
  Flanker Test of Attention (average reaction time on correct incongruent trials)
Response Inhibition | 18 weeks
  Percent correct on no-go trials on Go/No-Go Test
Working Memory | 18 weeks
  Average z-scores on two tests of working memory: 1)List Sorting Working Memory (total score which is the sum of scores on parts one and two) and Digit Span (sum of longest span forward and longest span backwards)
Verbal Memory | 18 weeks
  Logical Memory Story Recall (number of details correctly recalled on initial recall)
Speed of Processing | 18 weeks
  Digit Symbol Coding (number of correct responses in 60 seconds)
Cognitive Flexibility | 18 weeks
  Color/Word Stroop Test (Time to read words in conflicting colors minus time to read words without conflicting colors

CONTACTS AND LOCATIONS:
Overall Officials: Bruce E Wexler, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No